CLINICAL TRIAL: NCT03189875
Title: Systemic Lupus Erythematosus (SLE) Prospective Observational Cohort Study (SPOCS): Prospective Observational Cohort of Patients With Moderate-to-severe SLE to Characterize Cross-sectional and Longitudinal Disease Activity, Treatment Patterns and Effectiveness, Outcomes and Comorbidities, Healthcare Resource Utilization, and the Impact of SLE on Quality of Life by Type I Interferon Expression
Brief Title: Systemic Lupus Erythematosus (SLE) Prospective Observational Cohort Study (SPOCS)
Acronym: SPOCS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3461R00001
Record Dates: First submitted 2017-05-24; First posted 2017-06-16 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-01

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus Disease
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — type I IFN gene signature test (type 1 interferon gene test)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation: Cohort of patients with moderate-to-severe SLE
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Standard of Care — Participants will be followed as per local routine clinical practice

SUMMARY:
SPOCS is an international, multicenter, prospective observational cohort study with bi-annual study visits over a 3-year follow-up designed to systematically describe the comprehensive SLE patient-journey regarding clinical features, disease progression and treatment patterns, SLE outcomes, health status assessments (PROs), and health care resource utilization (HCRU) in a general population of moderate-to-severe SLE patients.

DETAILED DESCRIPTION:
SPOCS is an international, multicenter, prospective observational cohort study with bi-annual follow-up over 3-years maximum follow-up of patients with SLE confirmed by American College of Rheumatology (ACR) or Systemic Lupus International Collaborating Clinics (SLICC) classification criteria, who have moderate-to-severe disease by SLEDAI-2K criteria (Modified SLEDAI-2K score ≥4 and/or SLEDAI-2K score ≥6 points, at least one life-time positive serology of anti-nuclear antibody (ANA) or double-stranded deoxyribonucleic acid antibody (dsDNA), and 6-month minimum treatment duration with systemic SLE treatment beyond NSAIDS and analgesics. Participants will be followed as per local routine clinical practice. SPOCS is an observational study with no requirement for protocolized treatment interventions.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following criteria for enrollment in SPOCS:

* Adult patients aged 18 years or older
* Physician confirmation that patient meets ACR or SLICC SLE classification criteria
* Current or historic positive serology of ANA or dsDNA
* Minimum treatment duration of 6 months for active SLE with systemic SLE treatment beyond NSAIDs and analgesics
* Moderate-to-severe SLE; SLEDAI-2K Criteria: Modified SLEDAI-2K score ≥4 and/or SLEDAI-2K score ≥6. The "Modified" SLEDAI-2K is the SLEDAI-2K assessment score without the inclusion of points attributable to any urine or laboratory results including immunologic measures and lupus headache.
* Patient and/or representative(s) who understands the requirements of the study and provides written informed consent.

Exclusion Criteria:

Patients meeting any of the following criteria will be determined to be ineligible for enrollment in SPOCS:

* Patients actively enrolled in interventional trials involving investigational agents
* Patient with active severe lupus nephritis with a history of a renal biopsy in the last year showing active class III or class IV +/- class V lupus nephritis and/or urine protein:creatinine ratio >1mg/mg based on random urine collection.
* Patients unable to complete study measures

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of SLE confirmed by ACR or SLICC classification criteria with moderate-to-severe disease by SLEDAI-2K criteria (Modified SLEDAI-2K score ≥4 or SLEDAI-2K score ≥6 points), a historic or current positive serology for ANA or dsDNA, and a 6-month minimum treatment duration with systemic SLE treatment beyond NSAIDS and analgesics
Sampling Method: Non-Probability Sample
Enrollment: 830 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2022-11-18 (Actual)

PRIMARY OUTCOMES:
Disease activity | 6, 12, 18, 24, 30 and 36 months of follow-up
  Total Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score and score change from Baseline in patients with high and/or low status interferon 1 gene signature at Baseline after 6, 12, 18, 24, 30 and 36 months of follow-up.
Healthcare resource utilization including direct and indirect costs | 12, 24 and 36 months of follow-up
  Mean annual global healthcare cost related to SLE in patients with high and/or low status interferon 1 gene signature at Baseline after 12, 24 and 36 months of follow-up.
Patient reported health outcomes | 6, 12, 18, 24, 30 and 36 months of follow-up
  Total 36-Item Short Form Health Survey (SF-36) score and score change from Baseline in Physical Component Score (PCS) and Mental Component Score (MCS) in patients with high and/or low status interferon 1 gene signature after 6, 12, 18, 24, 30 and 36 months of follow-up. SF-36 survey covers eight domains of well-being: physical functioning, role limitations, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health combined into PCS and MCS, two summary scores of SF-36 survey.
Organ damage burden | 12, 24 and 36 months of follow-up
  Mean score for Systemic Lupus International Collaborating Clinics/American College of Rheumatology Damage Index (SLICC/ACR DI) and change from Baseline in SLICC/ACR DI for total score and individual components scores in patients with high and/or low status interferon 1 gene signature at Baseline after 12, 24 and 36 months of follow-up
Medical events of special interest | up to 36 months
  Incidence and prevalence of individual medical events of special interest in patients with high and/or low status interferon 1 gene signature at Baseline after 12, 24 and 36 months of follow-up.

CONTACTS AND LOCATIONS:
Locations (124):
- United States (30):
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Jonesboro, Arkansas
  - Research Site, Beverly Hills, California
  - Research Site, El Cajon, California
  - Research Site, Loma Linda, California
  - Research Site, Los Alamitos, California
  - Research Site, Los Angeles, California
  - Research Site, Mission Viejo, California
  - Research Site, San Francisco, California
  - Research Site, West Hills, California
  - Research Site, Miami, Florida
  - Research Site, Tamarac, Florida
  - Research Site, Coeur d'Alene, Idaho
  - Research Site, Chicago, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Baltimore, Maryland
  - Research Site, Detroit, Michigan
  - Research Site, Nashua, New Hampshire
  - Research Site, Newark, New Jersey
  - Research Site, Great Neck, New York
  - Research Site, The Bronx, New York
  - Research Site, Durham, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Salisbury, North Carolina
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Dallas, Texas
  - Research Site, The Woodlands, Texas
  - Research Site, Spokane, Washington
- Australia (10):
  - Research Site, Canberra, Australian Capital Territory
  - Research Site, Camperdown, New South Wales
  - Research Site, Liverpool, New South Wales
  - Research Site, New Lambton Heights, New South Wales
  - Research Site, Herston, Queensland
  - Research Site, Woodville South, South Australia
  - Research Site, Clayton, Victoria
  - Research Site, Fitzroy, Victoria
  - Research Site, Footscray, Victoria
  - Research Site, Nedlands, Western Australia
- Canada (13):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Halifax, Nova Scotia
  - Research Site, Barrie, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, London, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Ste-Foy, Quebec
- France (15):
  - Research Site, Strasbourg, Bas Rhin
  - Research Site, Caen, Calvados
  - Research Site, Corbeil-Essonnes, Essonne
  - Research Site, Bordeaux, Gironde
  - Research Site, Pessac, Gironde
  - Research Site, Montpellier, Herault
  - Research Site, Nantes, Loire Atlantique
  - Research Site, Cahors, Lot
  - Research Site, Angers, Maine Et Loire
  - Research Site, Vantoux, Moselle
  - Research Site, Lille, Nord
  - Research Site, Paris, Paris
  - Research Site, Lyon, Rhone
  - Research Site, Rouen, Seine Maritime
  - Research Site, Paris
- Germany (13):
  - Research Site, Heidelberg, Baden-Wurttemberg
  - Research Site, Stuttgart, Baden-Wurttemberg
  - Research Site, Munich, Bavaria
  - Research Site, Würzburg, Bavaria
  - Research Site, Bad Nauheim, Hesse
  - Research Site, Göttingen, Lower Saxony
  - Research Site, Bad Doberan, Mecklenburg-Vorpommern
  - Research Site, Wuppertal, North Rhine-Westphalia
  - Research Site, Ludwigshafen am Rhein, Rhineland-Palatinate
  - Research Site, Mainz, Rhineland-Palatinate
  - Research Site, Dresden, Saxony
  - Research Site, Berlin
  - Research Site, Dresden
- Italy (13):
  - Research Site, Monza, Milano
  - Research Site, Rozzano, Milano
  - Research Site, Rome, Roma
  - Research Site, Bologna
  - Research Site, Brescia
  - Research Site, Catania
  - Research Site, Florence
  - Research Site, Genova
  - Research Site, LAquila
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Pisa
  - Research Site, Torino
- Spain (13):
  - Research Site, Vitoria-Gasteiz, Alava
  - Research Site, L'Hospitalet de Llobregat, Barcelona
  - Research Site, Torrelavega, Cantabria
  - Research Site, El Palmar, Murcia
  - Research Site, Vigo, Pontevedra
  - Research Site, Oviedo, Principality of Asturias
  - Research Site, Bilbao, Vizcaya
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Granada
  - Research Site, Salamanca
  - Research Site, Seville
  - Research Site, Valladolid
- United Kingdom (17):
  - Research Site, Warrington, Cheshire
  - Research Site, Plymouth, Devon
  - Research Site, Brighton, East Sussex
  - Research Site, Eastbourne, East Sussex
  - Research Site, Harlow, Essex
  - Research Site, London, Greater London
  - Research Site, Maidstone, Kent
  - Research Site, Wigan, Lancashire
  - Research Site, Edinburgh, Lothian Region
  - Research Site, Liverpool, Merseyside
  - Research Site, Bath, Somerset
  - Research Site, Barnsley, South Yorkshire
  - Research Site, Doncaster, South Yorkshire
  - Research Site, Stoke-on-Trent, Staffordshire
  - Research Site, Coventry, Warwickshire
  - Research Site, Dudley, West Midlands
  - Research Site, Sheffield, West Midlands

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Morand EF, Furie R, Aringer M, Arnaud L, Peschken C, Hoi A, Lee KW, Hedberg J, Grunfeld Een T, Tummala R, Chen S, Ding B. Disease progression in patients with systemic lupus erythematosus: an analysis of the SLE Prospective Observational Cohort Study (SPOCS). Rheumatology (Oxford). 2025 Nov 11:keaf599. doi: 10.1093/rheumatology/keaf599. Online ahead of print. PMID 41217773
- [Derived] Aringer M, Arnaud L, Furie RA, Morand EF, Peschken C, Hoi A, Desta B, Hedberg J, Grunfeld Een T, Sorrentino A, Kielar D, Tummala R, Chen S, Ding B. Real-world treatment patterns and clinical characteristics in patients with moderate-to-severe systemic lupus erythematosus: an analysis of the SLE Prospective Observational Cohort Study (SPOCS). Lupus Sci Med. 2025 Jan 23;12(1):e001336. doi: 10.1136/lupus-2024-001336. PMID 39855677
- [Derived] Hammond ER, Tummala R, Berglind A, Syed F, Wang X, Desta B, Nab H. Study protocol for the international Systemic Lupus Erythematosus Prospective Observational Cohort Study (SPOCS): understanding lupus and the role of type I interferon gene signature. BMJ Open. 2020 Sep 1;10(9):e036563. doi: 10.1136/bmjopen-2019-036563. PMID 32873668
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3461R00001&attachmentIdentifier=365346ba-1f8d-495e-bc6b-76ac3abccb9d&fileName=SPOCS_CSR_Synopsis_Redacted.pdf&versionIdentifier=